CLINICAL TRIAL: NCT03770988
Title: A Single Arm Phase II Trial to Evaluate the Efficacy of Poziotinib, Pan HER Inhibitor in Recurrent/Metastatic Esophageal Cancer (R/M ESCC)
Brief Title: A Trial to Evaluate the Efficacy of Poziotinib, Pan HER Inhibitor in Recurrent/Metastatic Esophageal Cancer (R/M ESCC)
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 4-2017-1193
Record Dates: First submitted 2018-08-14; First posted 2018-12-10 (Actual); Last update posted 2019-02-22 (Actual); Status verified 2019-02

CONDITIONS: Inoperable or Recurrent or Metastatic Esophageal Squamous Carcinoma
Keywords: esophageal squamous carcinoma; poziotinib; pan-HER inhibitor
MeSH Terms: conditions — Recurrence | interventions — Therapeutics; HM781-36B

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- poziotinib single arm study (Experimental): Single Arm study
  Interventions: Drug: Treatment with Poziotinib

INTERVENTIONS:
Drug: Treatment with Poziotinib — Treatment with Poziotinib

SUMMARY:
Esophageal cancer is the sixth most common cause of cancer deaths worldwide. Esophageal adenocarcinoma has become more common in Western countries. In many Asian countries, however, Esophageal Squamous Cell Carcinoma (ESCC) represents the most common esophageal cancer. In palliative chemotherapy for metastatic or recurrent ESCC, A combination of 5-fluorouracil and platinum was prescribed as a standard treatment for about 20 years. With this traditional regimen, the median progression free survival is approximately 7 months, and 1-year survival rate is reported to be 34%. Combinations of taxane and anthracycline are also considerable, but also shows the median survival less than one year. Though cytotoxic chemotherapy is current main treatment option, molecularly targeted agents are recently incorporated to improve survival in ESCC. There is a strong rationale for investigation of biologic agents targeting Epithelial Growth Factor Receptor (EGFR) family in ESCC. EGFR is frequently overexpressed in esophageal cancer and is known to be associated with poor prognosis. Several EGFR tyrosine kinase inhibitors (TKIs) have been studied in esophageal cancer subjects and have shown clinical effects. In a recent Phase II trial using dacomitinib, pan-human epidermal growth receptor TKI, Partial response was observed in 10 of the 49 esophageal cancer subjects, with a response rate of 20.8%.

Based on notable rationale in exploring impact of EGFR inhibition, we suggest multicenter phase II study to determine antitumor activity and safety of a other potent pan-HER inhibitor, Poziotinib in Esophageal Squamous cell carcinoma.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically confirmed esophageal squamous cell carcinoma (Includes cases with pathologic findings with clinical course comparable to squamous cell carcinoma. For example, undifferentiated carcinoma)
2. Diseases that can not achieve curative aim with radical surgery, radiation, or chemo-radiotherapy. Previous palliative chemotherapy including platinum-based agents for advanced or recurrent esophageal squamous cell carcinoma (If the disease progresses within 6 months after the curative platinum-based chemotherapy or disease progresses within 6 months after last adjuvant chemotherapy, it is considered to be the previous palliative chemotherapy.
3. Have measurable disease based on RECIST 1.1.
4. Be 20 years of age on day of signing informed consent.
5. Performance status of 0 or 1 on the Eastern Cooperative Oncology Group Performance Scale.
6. Demonstrate adequate organ function
7. Absolute Neutrophil Count ≥ 1500/μL
8. Platelet Count ≥100,000/μL
9. Hemoglobin ≥ 9.0 g/dL
10. Serum creatinine ≤
11. Serum bilirubin ≤ 1.5 x ULN
12. AST, ALT ≤ 1.5 x ULN (with liver metastasis ≤ 5.0 x ULN)
13. Be willing and able to provide written informed consent/assent for the trial.

Exclusion Criteria:

1. Without measurable lesion based on RECIST 1.1
2. Has received prior therapy with EGFR/HER2 directed therapy.
3. Has history of intestinal obstruction or recent bleeding (subjects with clinically significant hemorrhagic or clotting events within the past 6 months)
4. Pregnant or lactating women
5. Women who have not received a baseline pregnancy test or have a positive result. (A woman who has not undergone a previous hysterectomy, or history of amenorrhea of more than 12 months, or undergone bilateral oophorectomy is considered to be a non-pregnant menopausal woman.)
6. Male or reproductive women who are not willing to use contraception during the trial
7. Has a known additional malignancy that is progressing or requires active treatment within 3 years. (Except skin basal cell carcinoma, cervix epithelial carcinoma in situ, Superficial bladder cancer)
8. Subjective who is likely to interfere with the understanding of the written consent or influence the compliance of the trial medication. Patients with a history of uncontrolled seizures, central nervous system disorders or psychiatric disorders that are considered clinically significant by the investigator
9. Has stable LVEF of less than 50%
10. Received organ transplants that require immunosuppressive therapy
11. Has un-controlled active infectious disease.
12. Has symptomatic central nerve system metastasis (Except in case of discontinuation of corticosteroids at least 2 weeks before clinical trials and radiologic and neurologically stable cases over 4 weeks)
13. Has known history of, or any evidence of active, non-infectious pneumonitis.
14. Has New York Heart Association, NYHA class III or IV Heart failure, un-controlled hypertension
15. Experienced unstable angina or myocardial infarction within the last 6 months
16. Has un-controlled arrhythmia or judged to have clinically significant cardiovascular abnormalities by investigators
17. Incapability of Oral ingestion and digestion.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 49 (Estimated)
Dates: Start 2019-04-01 (Estimated); Primary Completion 2020-08-31 (Estimated); Study Completion 2020-08-31 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate | every 8 weeks, assessed up to 100 weeks
  Objective Response Rate using RECIST 1.1

SECONDARY OUTCOMES:
Overall Survival | From date of randomization until date of death from any cause, whichever came first, assessed up to 100 months
Progression Free Survival | From date of randomization until date of death from any cause, whichever came first, assessed up to 100 months
Duration of Response | From date of randomization until date of death from any cause, whichever came first, assessed up to 100 months
Safety assessed by incidence of treatment-emergent adverse events | up to 100 weeks
  To evaluate the safety of Poziotinib, pan HER inhibitor in recurrent/metastatic esophageal cancer

CONTACTS AND LOCATIONS:
Locations (1):
- Severance Hospital, Seoul, South Korea